CLINICAL TRIAL: NCT01442051
Title: A Pilot Study of Acute Normovolemic Hemodilution in Patients Undergoing Cytoreductive Surgery for Advanced Ovarian Cancer
Brief Title: Acute Normovolemic Hemodilution in Patients Undergoing Cytoreductive Surgery for Advanced Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-149
Record Dates: First submitted 2011-09-23; First posted 2011-09-28 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2018-07

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: Acute Normovolemic Hemodilution; Cytoreductive Surgery; laparotomy; 11-149; advanced primary epithelial ovarian cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms

ARMS (1):
- Acute Normovolemic Hemodilution (Experimental): A pilot study will be performed. Intraoperative data including vital signs, procedures performed, and transfusions of allogenic blood will be collected prospectively. Postoperative outcomes, including transfusions of allogenic blood, perioperative complications, and 30-day mortality will be collected prospectively. These outcomes will be compared to historical controls to assess for the safety and efficacy of ANH in ovarian cancer cytoreductive surgery.
  Interventions: Procedure: Acute Normovolemic Hemodilution

INTERVENTIONS:
Procedure: Acute Normovolemic Hemodilution — A predetermined volume of whole blood will be removed from these patients based on an established protocol. Crystalloid and colloid will then be infused to replace intravascular volume based on this protocol. Patients will be closely monitored intraoperatively with serum arterial hemoglobin (HgB) levels drawn hourly. Patients will be transfused with autologous blood if HgB < 7.0 g/dL. If the volume of autologous blood has not been transfused within eight hours or by the completion of the procedure, the remainder will be transfused at that time. If the volume of autologous blood has been transfused and the patients require additional blood transfusions (HgB <7g.dL), allogenic blood will be transfused thereafter. These transfusion triggers are based on common intraoperative practice patterns. Patients may also be transfused intraoperatively at any time for a HgB ≥ 7.0 g/dL based on the judgment of the attending anesthesiologist or surgeon but the reason will be recorded.

SUMMARY:
The purpose of this study is to help us learn how to lower the risk of a blood transfusion during surgery to remove ovarian cancer. Acute normovolemic hemodilution (ANH) is a technique performed in the operating room before the procedure begins that may reduce the risk of needing a transfusion during ovarian cancer surgery. During surgery, the patient's own blood is given back to them when needed, usually due to bleeding. If you don't need blood during surgery, your own blood will be given back at the end of the case.

The idea behind ANH is that that by removing the blood and replacing it with other fluids, the remaining blood becomes diluted. This diluted blood is then lost during surgery, usually due to bleeding. The original non-diluted blood is then transfused back as needed. This may mean a lower chance of needing an additional blood transfusion.

ANH has been studied at this hospital for other types of cancer. These studies suggest that ANH may help conserve blood. Although most studies suggest that ANH can be performed safely, one study showed that ANH could be associated with a higher rate of serious bowel complications than standard treatment. In this study, patients who underwent ANH had a higher rate of anastomotic leaks during bowel surgery. An anastomotic leak occurs when two ends of bowel that have been cut and sewn back together (the anastomosis), fall apart. The investigators don't know whether ANH will result in higher rates of anastomotic leaks in patients having ovarian cancer surgery. In fact, in another study evaluating ANH in patients having the kind of bowel resections that often occur in ovarian cancer surgery (the colon), no increased risk of anastomotic leaks was observed. For these reasons, researchers at MSKCC are conducting a study to find out if ANH can be used safely in patients undergoing surgery for ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* The study population will include women with a high preoperative suspicion of advanced primary epithelial ovarian, fallopian tube, or primary peritoneal carcinoma (Stage IIIC or IV) as determined by CT or MRI of abdomen and pelvis planning to undergo exploratory laparotomy and surgical cytoreduction with the operative goal of this procedure to achieve optimal cytoreduction to less than 1 cm of residual disease.
* Age ≥ 18 years and < 70 years.
* Preoperative hemoglobin concentration ≥ 10 mg/dL within 30 days of registration.
* Based on surgeon's assessment, patient is recommended to undergo cytoreductive surgery via laparotomy with the operative goal of this procedure to achieve optimal cytoreduction to less than 1 cm of residual disease.

Exclusion Criteria:

* Hemoglobin < 10 g/dL.
* Serum albumin < 3g/dL.
* GOG performance status > 2.
* Active coronary artery disease (defined as unstable angina or a positive cardiac stress test).
* Patients with a history of coronary artery disease may be included if they have had a normal cardiac stress test within 30 days of enrollment.
* History of cerebrovascular disease.
* Renal insufficiency with serum creatinine > 1.6.
* Uncontrolled hypertension.
* Restrictive or obstructive pulmonary disease.
* Congestive heart failure.
* Active infection.
* Pregnancy.
* Refusal to accept allogenic or autologous blood transfusion.
* Autologous blood transfusion within last 30 days or plan to donate autologous blood prior to surgery.
* Plan for exploratory laparoscopy prior to laparotomy for assessment of disease resectability.
* Surgeon has high suspicion (>50% chance) that cytoreductive surgery will be aborted due to inability to achieve optimal cytoreduction to < 1cm residual disease.

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-09-23 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
the safety of performing acute normovolemic hemodilution (ANH) | within 7 days
  Allogenic red blood cell transfusion rate will be measured as any transfusion during the operating procedure or during the hospitalization

SECONDARY OUTCOMES:
impact on transfusion rates | 2 years
  Allogenic red blood cell transfusion rate will be measured as any transfusion during the operating procedure or during the hospitalization. The charts of patients transfused outside of the guidelines will be flagged for auditing and will be reviewed by the PI. Such transfusions will be considered appropriate if a reasonable clinical justification is identified.
length of hospitalization stay | 2 years
postoperative complications | within 30 days of surgery
  Careful assessment and recording of all intraoperative and postoperative complications within 30 days of surgery according to universal guidelines as established by the Gynecologic Oncology Group and affirmed by the Division of Gynecology at MSKCC.
operating time | Duration of surgical procedure
  operative time will be compared to historical controls that received standard intraoperative management.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Chi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm